CLINICAL TRIAL: NCT04563455
Title: Investigation of the Relationship Between Grip Endurance, Disability of Upper Extremity and Quality of Life in Patients With Rheumatoid Arthritis
Brief Title: Relationship Between Grip Endurance, Disability of Upper Extremity and Quality of Life in Patients With RA
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Melissa Köprülüoğlu, Research Assistant, Izmir Katip Celebi University
Other Study IDs: IzmirKatip Celebi University
Record Dates: First submitted 2020-09-23; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Grip Endurance, DASH, Quality of Life, Rheumatoid Arthritis.
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the relationship between grip endurance, disability of upper extremity and quality of life in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Upper extremity functions affect the quality of life at different levels in patients with rheumatoid arthritis (RA). In the current literature; it has been shown that grip endurance is associated with upper limb functions. However, there is no study investigating the relationship between grip endurance and quality of life in patients with RA. The purpose of this study is to investigate the relationship between grip endurance, disability of upper extremity, and quality of life in patients with RA.

ELIGIBILITY:
Inclusion Criteria:

* RA patients were classified according to the ACR 2010 criteria.
* taking regular medication.

Exclusion Criteria:

* having a history of trauma or surgery in the upper limb.
* having neurological, cognitive, or psychiatric diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study consists of RA patients.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Static Grip Endurance | Data collection will continue until December 2019. Data analysis and report preparation will be completed by September 2020.
  Static grip endurance was evaluated by Hand Dynamometer (Lafayette Proffessional Hand Dynamometer, USA). The maximum gripping time of 50% of the maximum grip force was recorded.
Dynamic Grip Endurance | Data collection will continue until December 2019. Data analysis and report preparation will be completed by September 2020.
  Dynamic grip endurance was evaluated by Hand Dynamometer (Lafayette Proffessional Hand Dynamometer, USA). The percentage change between the first 3 grips and the last 3 grips after 10 consecutive grips is recorded.

SECONDARY OUTCOMES:
Disability of Upper Extremity | Data collection will continue until December 2019. Data analysis and report preparation will be completed by September 2020.
  This parameter was evaluated by Disability of Arm, Shoulder and Hand (DASH) questionairre.
Quality of Life Parameters | Data collection will continue until December 2019. Data analysis and report preparation will be completed by September 2020.
  This parameter was evaluated by Short Form-36.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa KÖPRÜLÜOĞLU, Principal Investigator — İzmir Katip Celebi University, Faculty of Health Sciences
Locations (1):
- Izmir Katip Celebi University, Izmir, Izmir/ Cigli, Turkey (Türkiye)